CLINICAL TRIAL: NCT01085955
Title: Immune Activation and Myocardial Recovery in Peripartum Cardiomyopathy
Brief Title: Investigation in Pregnancy Associate Cardiomyopathy
Acronym: IPAC
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Dennis McNamara, Prinicipal Investigator, University of Pittsburgh
Other Study IDs: IPAC
Record Dates: First submitted 2010-03-10; First posted 2010-03-12 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Cardiomyopathy; Pregnancy
Keywords: peripartum; cardiomyopathy; post pregnancy; myocardial recovery; pregnant women with peripartum cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens for cellular analysis, complete blood count, DNA banking and genotyping, RNA analysis and banking, serum banking and for mediator analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Acute Peripartum: pregnant women who have recently given birth and diagnosed with peripartum cardiomyopathy
- Healthy Peripartum: Healthy pregnant women who have recently given birth, used as controls
- Healthy, non-pregnant women: Healthy non-pregnant women without cardiac disease, used as controls
- New Non-ischemic CMP: Women 18-60 years old who have been diagnosed with non-ishemic cardiomyopathy within the last 6 months and have an ejection fraction less than OR equal to 45% by echocardiogram.

SUMMARY:
Peri-partum cardiomyopathy is a heart muscle weakness that occurs during or following pregnancy. Research suggests that many initial heart injuries including viruses, pregnancy and other unknown causes, can lead to a process of inflammation of the heart muscle which can weaken the heart and cause cardiomyopathy. Why this process occurs in women during pregnancy is not well understood and if it differs from those women who develop cardiomyopathy from a virus is unknown. This study has been proposed to look at genetic information (DNA) as well as the immune system (the body's response to fight off infections and/or viruses) to find possible causes for the heart muscle damage that occurs in peripartum cardiomyopathy.

DETAILED DESCRIPTION:
Specific Aim 1: Evaluate systemic immune activation as the etiology of PPCM. We will determine a) the degree of immune activation in PPCM and b) the relationship of autoimmunity to left ventricular dysfunction and time course of myocardial recovery, in 100 women enrolled at 30 centers. Subjects will have blood drawn for assessment of autoantibodies, and cellular immune activation at presentation, 2 month and 6 month postpartum, and will have assessment of LVEF by transthoracic echo at presentation, 2 months, 6 months and 12 months post partum. This aim will explore the hypothesis that more prolonged activation of the cellular and/or humoral immune system is associated with greater likelihood of persistent chronic cardiomyopathy.

In addition this aim will determine genetic and clinical predictors of LV recovery, and evaluate racial differences in presentation, remodeling and recovery. This study will evaluate the echo parameters of dysynchrony, diastolic function, LV size and volumes to determine echo predictors of subsequent recovery. In addition racial differences in presentation, remodeling and recovery will be investigated.

Specific Aim 2: Investigate frequency of myocardial injury or inflammation on cardiac MRI and the ability of tissue characteristics to predict subsequent recovery of LVEF. Cardiac MRI with gadolinium enhancement will be performed in 50 subjects with PPCM from Aim 1 at presentation and repeated at 6 months post partum. We will test the hypothesis is that subjects with more extensive injury (defined as % myocardium with late gadolinium enhancement) will have less recovery at 6 months.

Specific Aim 3: Establish DNA and serum to facilitate future investigations of the pathogenesis of peripartum cardiomyopathy. All subjects enrolled will have DNA, RNA from peripheral blood and serum banked at entry. Serum will be repeated at 2 and 6 months post partum.

ELIGIBILITY:
Inclusion Criteria:

* Patient of 16 years of age or older
* Diagnosis of peripartum cardiomyopathy
* Presentation for enrollment no earlier than one month pre-term and no later than two months post partum.
* LVEF less than OR equal to 0.45 by echocardiogram

Additional inclusion criteria for MRI substudy:

* Must be post partum
* Participant is not breast feeding or is willing to forego breast feeding for 24 hours post gadolinium.

Exclusion Criteria:

* Previous diagnosis of cardiomyopathy, valvular disease or complex congenital heart disease
* Evidence of CAD (>50% stenosis of major epicardial vessel or positive non-invasive stress test)
* Previous cardiac transplant
* Chemotherapy or chest radiation within 5 years of enrollment
* Evidence of ongoing bacterial septicemia (positive blood cultures)
* Medical, social, or psychiatric condition which limit the ability to comply with follow-up (Example: alcohol or drug abuse)

Additional Exclusion for MRI Substudy

* GFR < 30mL/1.7 m2 by MDRD equation (http://www.kidney.org/professionals/kdogi/gfr_calculator.cfm)
* Currently breast feeding or unwilling to forego for 24 hour period post gadolinium
* Implanted devices (cochlear implants, pacemakers, defibrillators, infusion pumps, nerve stimulators, etc)
* Cerebral aneurysm clips
* Swan Ganz catheter or intra aortic balloon pump
* Ocular metal or metallic splinters in the eye
* Pregnant women
* Metal shrapnel or bullet
* Allergy to Gadolinium

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 100 women diagnosed with peripartum cardiomyopathy
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Evaluate systemic immune activation as the etiology of PPCM | 6-12 months
  determine the degree of immune activation in PPCM and the relationship of autoimmunity to left ventricular dysfunction and time course of myocardial recovery, in 100 women enrolled at multiple centers.

SECONDARY OUTCOMES:
Investigate frequency of myocardial injury or inflammation on cardiac MRI and the ability of tissue characteristics to predict subsequent recovery of LVEF | 6 months
  Cardiac MRI with gadolinium enhancement will be performed in 50 subjects with PPCM from Aim 1 at presentation and repeated at 6 months post partum. We will test the hypothes that subjects with more extensive injury (defined as % myocardium with late gadolinium enhancement) will have less recovery at 6 months

OTHER OUTCOMES:
Long Term Survival Data | up to 5 years
  We are asking women to extend thier consent for 5 additional years from thier delivery date to collect survival data (alive, transplanted, VAD implanted; medications; NYAH Class; subsequent pregnancies)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis McNamara, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (30):
- United States (28):
  - University of Southern California, Los Angeles, California
  - University of Miami, Miller School of Medicine, Miami, Florida
  - Medical College of Georgia, Augusta, Georgia
  - University of Illinois, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Louisiana State University Health Science Center, Louisiana, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General, Boston, Massachusetts
  - Brigham and Women's, Boston, Massachusetts
  - DMC Cardiovascular Institute / Harper University Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Gagnon Cardiovascular Institute at Morristown Memorial Hospital, Morristown, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Duke University, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas, Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
- Canada (2):
  - Foothills Medical Center, Calgary, Alberta
  - Sir Mortimer B. Davis / Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Schelbert EB, Elkayam U, Cooper LT, Givertz MM, Alexis JD, Briller J, Felker GM, Chaparro S, Kealey A, Pisarcik J, Fett JD, McNamara DM; Investigations of Pregnancy Associated Cardiomyopathy (IPAC) Investigators. Myocardial Damage Detected by Late Gadolinium Enhancement Cardiac Magnetic Resonance Is Uncommon in Peripartum Cardiomyopathy. J Am Heart Assoc. 2017 Apr 3;6(4):e005472. doi: 10.1161/JAHA.117.005472. PMID 28373243
- [Derived] Damp J, Givertz MM, Semigran M, Alharethi R, Ewald G, Felker GM, Bozkurt B, Boehmer J, Haythe J, Skopicki H, Hanley-Yanez K, Pisarcik J, Halder I, Gorcsan J 3rd, Rana S, Arany Z, Fett JD, McNamara DM; IPAC Investigators. Relaxin-2 and Soluble Flt1 Levels in Peripartum Cardiomyopathy: Results of the Multicenter IPAC Study. JACC Heart Fail. 2016 May;4(5):380-8. doi: 10.1016/j.jchf.2016.01.004. Epub 2016 Mar 9. PMID 26970832
- [Derived] McNamara DM, Elkayam U, Alharethi R, Damp J, Hsich E, Ewald G, Modi K, Alexis JD, Ramani GV, Semigran MJ, Haythe J, Markham DW, Marek J, Gorcsan J 3rd, Wu WC, Lin Y, Halder I, Pisarcik J, Cooper LT, Fett JD; IPAC Investigators. Clinical Outcomes for Peripartum Cardiomyopathy in North America: Results of the IPAC Study (Investigations of Pregnancy-Associated Cardiomyopathy). J Am Coll Cardiol. 2015 Aug 25;66(8):905-14. doi: 10.1016/j.jacc.2015.06.1309. PMID 26293760